CLINICAL TRIAL: NCT03669653
Title: Safety and Efficacy of Remote Ischemic Conditioning in Patients With Acute Ischemic Stroke
Acronym: SERIC-AIS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yi Yang (Other)
Responsible Party: Sponsor-Investigator, Yi Yang, Clinical Trial and Research Center for Stroke, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SERIC-AIS
Record Dates: First submitted 2018-08-27; First posted 2018-09-13 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-02

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIC+Standard medical treatment (Active Comparator): Remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min reperfusion. Limb ischemia was induced by inflations of a blood pressure cuff to 200 mm Hg. RIC will be conducted twice daily for 7 days. Additionally,the patients will be treated with standard medical treatment according to Guidelines for diagnosis and treatment of acute ischemic stroke in China 2014
  Interventions: Procedure: Remote ischemic conditioning
- Sham RIC+Standard medical treatment (Placebo Comparator): Remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min reperfusion. Limb ischemia was induced by inflations of a blood pressure cuff to 60 mm Hg. RIC will be conducted twice daily for 7 days. Additionally,the patients will be treated with standard medical treatment according to Guidelines for diagnosis and treatment of acute ischemic stroke in China 2014
  Interventions: Procedure: Sham remote ischemic conditioning

INTERVENTIONS:
Procedure: Remote ischemic conditioning — Remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min reperfusion. Limb ischemia was induced by inflations of a blood pressure cuff to 200 mm Hg. RIC will be conducted twice daily for 7 days.
  Arms: RIC+Standard medical treatment
Procedure: Sham remote ischemic conditioning — Remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min reperfusion. Limb ischemia was induced by inflations of a blood pressure cuff to 60 mm Hg. RIC will be conducted twice daily for 7 days.
  Arms: Sham RIC+Standard medical treatment

SUMMARY:
he purpose of this study is to determine the efficacy and safety of remote ischemic conditioning for acute ischemic stroke.

DETAILED DESCRIPTION:
In this study, 912 cases of ischemic stroke in 48 hours were included in 5 centers in China according to the principle of random, double-blind and parallel control .The experimental group receive basic treatment and remote ischemic conditioning for 200mmHg, 2 times per day for 7 consecutive days .The control group receive basic treatment and remote ischemic conditioning control for 60mmHg, 2 times per day, 7 days in a row . Two groups will be followed up for 90 days to evaluate the efficacy and safety of remote ischemic conditioning therapy.

ELIGIBILITY:
Inclusion Criteria:

* 1）Age≥18 years, < 80 years, regardless of sex；
* 2）Patients with clinically definite diagnosis of acute ischemic stroke and able to commence RIC treatment within 12 hours of stroke onset
* 3）Baseline NIHSS score>5, and≤25 ；
* 4）GCS score ≥8；
* 5）Signed and dated informed consent is obtained

Exclusion Criteria:

* 1) Patients with suspected posterior circulation infarction；
* 2) Patients who undergo thrombolytic therapy or endovascular treatment；
* 3) mRS≥2 score before the onset of the disease；
* 4) Double upper limbs or lower limbs paralysis was found in this case；
* 5）Active bleeding of organs within 6 months of admission or current, including cerebral hemorrhage, subarachnoid hemorrhage, gastrointestinal hemorrhage, fundus hemorrhage and so on；
* 6) Other intracranial lesions, such as cerebrovascular malformation cerebral venous diseases, tumor and other diseases involving the brain；
* 7) Treated blood pressure ≤90mmHg/60mmHg or≥180mmHg/100mmHg；
* 8) Severe organ dysfunction or failure；
* 9) Persons suffering from severe hematological diseases or severe coagulation disorder dysfunction；
* 10) Those who had a history of severe trauma or had major surgery within 6 months prior to admission；
* 11) The patients who had the contraindication of remote ischemic conditioning treatment, such as severe soft tissue injury, fracture or vascular injury in the upper limb；Acute or subacute venous thrombosis, arterial occlusive disease, subclavian steal syndrome, etc；
* 12) Pregnant or lactating women；
* 13) Previous remote ischemic conditioning therapy or similar treatment；
* 14) Patients with a life expectancy of less than 3 months or patients unable to complete the study for other reasons；
* 15) Severe hepatic and renal dysfunction
* 16) Unwilling to be followed up or treated for poor compliance；
* 17) He/She is participating in other clinical research or has participated in other clinical research or has participated in this study within 3 months prior to admission；
* 18) Other conditions that the researchers think are not suitable for the group.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 912 (Estimated)
Dates: Start 2025-06-17 (Estimated); Primary Completion 2026-09-20 (Estimated); Study Completion 2026-09-20 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with Modified Rankin Scale (mRS) Score 0-2 | 3 months
  The primary outcome measure of efficacy is the modified Rankin Scale (mRS) dichotomized to define good functional outcome as mRS 0-2 at 90 days.score, dichotomized to define good functional outcome as mRS 0-2 at 90 days.

SECONDARY OUTCOMES:
NIHSS Score at end of 7th day of treatment | 7 days
  NIHSS Score at end of 7th day of treatment
mRS Score at end of 7th day of treatment | 7 days
  mRS Score at end of 7th day of treatment
Barthel Index at end of 7th day of treatment | 7 days
  Barthel Index at end of 7th day of treatment
Changes of hematological indicators | 48h; 7days
  The changes of hematological indicators (inflammatory cytokine,et al.) between the first 48h and end of 7th day of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China